CLINICAL TRIAL: NCT02526381
Title: Study on the Relation Between Syndrome and Disease of Turbid Phlegm and Blood Stasis for Coronary Heart Disease and Its Biological Basis
Brief Title: Clinical Study On The Relation Among Prescription, Syndrome and Disease of Turbid Phlegm and Blood Stasis for Coronary Heart Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tianjin University of Traditional Chinese Medicine (Other)
Responsible Party: Principal Investigator, Chunquan Yu, Director,Clinical Research, Tianjin University of Traditional Chinese Medicine
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: 2014CB542902
Record Dates: First submitted 2015-08-14; First posted 2015-08-18 (Estimated); Last update posted 2015-11-20 (Estimated); Status verified 2015-11

CONDITIONS: Coronary Heart Disease
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Danlou Tablets (Experimental): Danlou prescription is a tablet, each piece weighs 0.3 g, taken orally, three times a day, five at a time, from jilin Cornell's pharmaceutical corporation, Limited Liability Company .
  Interventions: Drug: Danlou Tablets
- Tongmai Yangxin Pills (Experimental): Tongmai Yangxin prescription is a pill,each pill weighs 0.1 g,taken orally, 2 times a day,40 pills at a time,produced by tianjin new pharmaceutical group corporation, Limited Liability Company . LeRenTang pharmaceutical.
  Interventions: Drug: Tongmai Yangxin Pills
- no drugs (No Intervention)

INTERVENTIONS:
Drug: Danlou Tablets — Five tablets of Danlou Tablets (1.5g) will be given three times a day in addition to regular western medications for the 8 weeks
  Arms: Danlou Tablets
Drug: Tongmai Yangxin Pills — Forty pills of Tongmai Yangxin Pills (4g) will be given two times a day in addition to regular western medications for the 8 weeks
  Arms: Tongmai Yangxin Pills

SUMMARY:
Clinical study on patients with turbid phlegm and blood stasis syndrome and Qi -Yin Deficiency syndrome of coronary artery disease (CHD) compared with normal cases will be launched. Detection of lipid metabolism, inflammation medium, endothelial cell injury, blood coagulation function evaluation of the relationship between disease and biochemical basis, detect plasma metabonomics and the gene expression profile chip, with "phlegm - lipid metabolic disorder", "stasis - microcirculation disorder", "alternating knot - inflammation mediated" and other system related to the biological basis. With Danlou Tablet for treatment, the investigators can observe result/effect index of turbid phlegm and blood stasis syndrome. Through comprehensive comparison of multi-level, multi-targets and multi-date biological index to discuss its sickness-syndrome-prescription corresponding relation and its biological basis.

ELIGIBILITY:
Inclusion Criteria:

1. Selecting people aged between 35 and 65;
2. Being up to the western diagnostic standard of chronic stable angina(complying with one or more of the following ): 1) There is a clear history of old myocardial infarction; 2) Have undergone coronary angiography or coronary Computed Tomography angiography(CTA) inspection hint antrum of coronary artery with at least a major branch pipe diameter stenosis≥50%; 3) Have received percutaneous coronary intervention (PCI) or Coronary Artery Bypass Grafting(CABG) treatment.
3. They should sign the informed consent.

Exclusion Criteria:

1. Had history of myocardial infarction or unstable angina, or coronary artery revascularization in 3 months.(coronary artery bypass graft or angioplasty);
2. With other diseases that might cause chest pain, including heart diseases, neurosis, menopausal syndrome,hyperthyroidism, Cervical vertebra sickness (arteria vertebrals and spinal cord), gastroesophageal reflux disease or hiatal hernia.
3. Using three or more of these drugs,namely beta blockers, calcium channel blockers, Energy metabolism drugs，and nitrate medications;
4. With hypertension and blood pressure after Anti-hypertensive Medical Therapy is still on the high side (systolic pressure ≥160 mmHg,diastolic pressure ≥100 mmHg)combined with severe cardiopulmonary insufficiency or severe arrhythmia (Rapid auricular fibrillation, atrial flutter or Paroxysmal Supra VentricularTachycardia);
5. Having liver disease or with unexplained serum transaminase continually increasing, or alanine aminotransferase(ALT) and aspartate aminotransferase (AST) greater than 2-fold of the upper limit of normal reference value;
6. Abnormal renal function;
7. Merger of hematopoietic system diseases, or a serious primary diseases such as malignant tumor;
8. Pregnant women, nursing mothers, or there is a requirement for fertility of women of childbearing age;
9. Diabetic kidney disease, severe gouty nephropathy and other metabolic diseases;
10. People with severe metabolic disease;
11. People who are expected with poor medical compliance or can't be visited on a regular basis;
12. Have participated in other clinical trials in recent 3 months;
13. Researchers considering there are other cases in which people are not suitable for attending the trial.

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2015-07; Primary Completion 2017-12 (Estimated); Study Completion 2018-08 (Estimated)

PRIMARY OUTCOMES:
Traditional Chinese Medicine symptom scores of Turbid Phlegm and Blood Stasis for Coronary Heart Disease | 12 weeks
Seattle Angina Questionnaire | 12 weeks
The Short Form (36) Health Survey, (SF-36) | 12 weeks
Self-reporting Inventory(symptom checklist-90) | 12 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin University of Traditional Chinese Medicine, Tianjin, Tianjin Municipality, China